CLINICAL TRIAL: NCT04187846
Title: Evaluation of the Relationship Between Postspinal Headache and Near Infrared Spectroscopy in Cesarean Section Patients
Brief Title: Postspinal Headache and Near Infrared Spectroscopy (NIRS)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hakan Tapar (Other)
Responsible Party: Sponsor-Investigator, Hakan Tapar, Assistant professor, Tokat Gaziosmanpasa University
Organization: Tokat Gaziosmanpasa University (Other)
Other Study IDs: 18-KAEK-167
Record Dates: First submitted 2019-12-02; First posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Tissue Oxygenation
Keywords: Cesarean section; post spinal headache; Near Infrared spectroscopy
MeSH Terms: conditions — Post-Dural Puncture Headache

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of the relationship between postspinal headache and near infrared spectroscopy in cesarean section patients

DETAILED DESCRIPTION:
Patients with cesarean section under spinal anesthesia were included in the study. Before the study, patients were moniterized with NIRS device in the preoperative waiting room.NIRS moniterization was continued intraoperatively at 1st, 4th, 7th, 10th, 15th, 30th minutes and 24th postoperative period.

Patients were divided into two groups as those with postspinal headache (Group A) and those with postspinal headache (Group B). In this study, NIRS values between two groups were compared.

ELIGIBILITY:
Inclusion Criteria:

* Elective cesarean section

Exclusion Criteria:

* Not willing to participate in the study
* Use of anti-psychotic or anti-depressant drugs
* Patients with headaches

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with cesarean section under spinal anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-03-10 (Estimated)

PRIMARY OUTCOMES:
Near Infrared spectroscopy | Up to 20 weeks
  Tissue oxygenation

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Tapar, Principal Investigator — Gaziosmanpasa University
Locations (1):
- Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)